CLINICAL TRIAL: NCT00911209
Title: Impact of Weight Loss on Diastolic Dysfunction in Overweight Pre-Hypertensives
Brief Title: Weight Loss in Pre-Hypertensive Patients With Diastolic Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated because funding was not found
Sponsor: Ragavendra Baliga (Other)
Responsible Party: Sponsor-Investigator, Ragavendra Baliga, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007H0328
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Heart Disease; Weight Loss; Diastolic Dysfunction
Keywords: Heart Disease; Obesity
MeSH Terms: conditions — Obesity; Heart Diseases; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The Intervention group at each session will receive information on Heart healthy diet, lifestyle recommendations and diet and exercise counseling with a dietitian in order to achieve at least 7% weight loss (for example a person weighing 200 pounds will be encourage to lose at least 14 pounds).
  Interventions: Behavioral: Dietitian counselling
- No Intervention (No Intervention): The standard of care group will receive information on Heart healthy diet at baseline visit and will return to a final visit about 28 weeks later.

INTERVENTIONS:
Behavioral: Dietitian counselling — Once a week for 14 weeks then 1 monthly visit. Visits last 40-50 minutes
  Arms: Intervention

SUMMARY:
The focus of this study is to observe the impact of weight loss in overweight individuals who have pre-hypertension (have a blood pressure reading of 121-139/81-89 mm Hg). The specific focus is to observe the difference in diastolic dysfunction (heart function) in these individuals at the beginning of the study and then again after 24-28 weeks. Diastolic dysfunction in this population indicates an increased risk of heart failure in the future. The aim of this study is to prevent or reduce the risk of heart failure in overweight individuals with pre-hypertension.

DETAILED DESCRIPTION:
You will be enrolled in the study for 24-28 weeks and will be randomly assigned to one of two assigned group. One group of subjects (Intervention group) will receive information on Heart healthy diet, lifestyle recommendations and diet and exercise counseling with a dietitian in order to achieve at least 7% weight loss. The other group will receive standard of care i.e., Information on Heart healthy diet at baseline visit (Standard of care group). The following is the time line of activities anticipated by the subject in each group. Both the groups will be screened at 3 different visits within 4 weeks to determine eligibility. If you are eligible they will be randomized to either be in Standard of care group or Intervention group. After randomization, the "Standard of care group" will come for Baseline and Final visit (24th week). The Intervention group will have 14 weekly visits with a nutritionist and 1 monthly visit, about 40-50 minutes each visit (total of 15) in 24- 28 week time frame. The second monthly session will be the final assessment visit. Both the groups will have a Baseline Assessment and a Final Assessment visit which will last about 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 21 years
* BMI ≥30
* Individuals with diagnosis pre-hypertension at the time of screening, defined as either a blood pressure measurement of 130-139/85-89 mm Hg
* Echocardiographic EF >50%
* Echocardiographic evidence of diastolic dysfunction;

Exclusion Criteria:

* Patients receiving antihypertensive medications
* Patients receiving diabetic medication

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Determine if weight loss is associated with changes in separate components of cardiac function. | 32 weeks

SECONDARY OUTCOMES:
Determine whether specific cardiac markers will be altered in patients with diastolic dysfunction treated with low caloric diet and exercise and if these levels will be altered in association with improvement in diastolic function. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ragavendra Baliga, MD, MBA,, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States